CLINICAL TRIAL: NCT07097792
Title: Pilot Study of Concussion Recovery and Support Program (CRISP)
Brief Title: Concussion Recovery and Support Program
Acronym: CRISP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Sara PD Chrisman, MD MPH, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00005446
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Brain Concussion; Mild Traumatic Brain Injury; Headache
Keywords: mental health; therapy; emotional awareness and expression therapy
MeSH Terms: conditions — Brain Concussion; Headache; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Data analyst will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRISP (Experimental): CRISP is an adaptation of an approach called EAET that was originally designed to treat individuals with chronic pain. The goal of this approach is to target underlying emotional reactions that may be causing symptoms to persist. This intervention will be delivered in 6 sessions over 10 weeks.
  Interventions: Behavioral: CRISP (Concussion Recovery and Support Program)
- Treatment as usual (TAU) (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: CRISP (Concussion Recovery and Support Program) — Mental health intervention targeting suppressed emotion with a goal of facilitating recovery.
  Arms: CRISP

SUMMARY:
Pilot randomized controlled trial (RCT) comparing a novel intervention Concussion Recovery and Support Program (CRISP) for adolescents and young adults (AYA) 18-29 yo with concussion/ mild TBI.

DETAILED DESCRIPTION:
The authors are conducting a pilot study to examine the feasibility, acceptability and pilot efficacy of a novel intervention called CRISP for young adults with persistent concussion/ mTBI. CRISP is an adaptation of an evidence-based treatment for chronic pain called Emotional Awareness and Expression Therapy (EAET). EAET targets underlying emotional responses that appear to drive persistent symptoms, and has been found effective for treating headache and other types of pain in randomized controlled trials with moderately strong effect sizes (0.4-0.5).

Individuals who participate in this study will complete 6 sessions of CRISP with a trained therapist over zoom (each 60 minutes) and will also fill out surveys at multiple time points (baseline, 5 weeks, 10 weeks).

Aim 1: Evaluate feasibility and acceptability of CRISP with a pilot study of n=40 individuals with concussion ages 18-30 years who are struggling with headache. Hypothesis: CRISP will be a feasible and acceptable approach to treating AYA with concussion.

Aim 2: Collect pilot data regarding efficacy of CRISP for reducing concussion symptoms and improving function (particularly regarding headache). Hypothesis: Pilot data may show benefit from this approach for improving recovery, though we do not expect significance given the sample size.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a concussion and at least 2 weeks from injury but less than two years.
* New or worsening headache since concussion
* Had at least one day with headache last week of moderate severity or two days with headache of any severity

Exclusion Criteria:

* Non-English speaking
* Chronic medical illness/ medical complexity
* Housing instability
* Acute mental health issues such as active suicidality, psychiatric hospitalization within the past 6 months, ER visit for suicidality in the past 6 months or experiencing psychosis or delusions

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Evaluation Inventory, short form | 10 weeks
  Self-report form regarding acceptability of treatment approach. Minimum 0, maximum 24 (6 items x 4 likert), higher scores indicate higher rating of treatment acceptability.

SECONDARY OUTCOMES:
HIT6 (Headache Impact Test, 6 item) | Baseline, 5 weeks, 10 weeks (trajectory over time)
  Self-report measure of headache severity, minimum 6 maximum 78, higher scores indicates greater symptoms.
PROMIS fatigue short form | Baseline/ 5 weeks/ 10 weeks (trajectory over time)
  7 item self-report scale measuring issues with fatigue. Minimum 7, maximum 35, higher scores indicates more symptoms.
Fear of Concussive Symptoms Questionnaire (FOCSQ) | Baseline/ 5 weeks/ 10 weeks (trajectory over time)
  Self-report measure of fear-avoidance of activities due to concussive symptoms. Minimum 0, maximum 96 (24 items x 4 likert), higher is worse
Post Concussion Symptom Scale (PCSS) | Baseline/ 5 weeks/ 10 weeks (trajectory over time)
  Self-report measure of concussive symptoms, minimum 0, maximum 132 (22 items x 6 likert), higher indicates more symptoms
PROMIS (Patient Reported Outcome Measurement Information System) anxiety | Baseline/ 5 weeks/ 10 weeks (trajectory over time)
  8 item scale to measure self-report of anxiety, minimum 8, maximum 40 (5likert x 8), higher indicates more symptoms
PROMIS depression | Baseline/ 5 weeks/ 10 weeks (trajectory over time)
  8 item scale to measure self-report of depressive symptoms, minimum 8, maximum 40 (5 likert x 8 items), higher indicates more symptoms
Emotional Approach Coping (EAC) | Baseline/ 5 weeks/ 10 weeks (trajectory over time)
  Self-report survey to measure ability to acknowledge and express emotion, minimum 8, maximum 32 (4 likert x 8), higher indicates more symptoms
Psychological Insight | 10 weeks (post-intervention only)
  6 item self-report scale to measure psychological insight, minimum 0, maximum 24 (4 likert x 6), higher indicates greater insight
PROMIS sleep disturbance SF | Baseline/ 4 weeks/ 8 weeks (trajectory over time)
  Self-report measure of sleep disturbance, minimum 8, maximum 40 (5 likert x 8), higher indicates more symptoms

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Seattle Children's Research Institute, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Would consider sharing in a collaborative fashion given pilot nature of study

REFERENCES:
- [Background] Lumley MA, Schubiner H. Emotional Awareness and Expression Therapy for Chronic Pain: Rationale, Principles and Techniques, Evidence, and Critical Review. Curr Rheumatol Rep. 2019 May 23;21(7):30. doi: 10.1007/s11926-019-0829-6. PMID 31123837